CLINICAL TRIAL: NCT07019636
Title: Direct Extubation Versus Extubation After a Spontaneous Breathing Trial in Patients at Low Risk of Extubation Failure
Acronym: T-REX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP240912; 2025-A00258-41 (Other: ANSM)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Weaning From Mechanical Ventilation, Extubation
Keywords: Weaning; Mechanical ventilation; Extubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weaning strategy with direct extubation (no spontaneous breathing trial) (Experimental)
  Interventions: Procedure: Weaning strategy with direct extubation (no spontaneous breathing trial)
- Weaning strategy with extubation only after a successful spontaneous breathing (Active Comparator)
  Interventions: Procedure: Weaning strategy with extubation only after a successful spontaneous breathing

INTERVENTIONS:
Procedure: Weaning strategy with direct extubation (no spontaneous breathing trial) — Patients will be extubated within the 60 minutes following randomization
  Arms: Weaning strategy with direct extubation (no spontaneous breathing trial)
Procedure: Weaning strategy with extubation only after a successful spontaneous breathing — Patients will undergo a spontaneous breathing trial and will be extubated only in case of successful spontaneous breathing
  Arms: Weaning strategy with extubation only after a successful spontaneous breathing

SUMMARY:
This randomized controlled open label trial aims at comparing a weaning strategy including a spontaneous breathing trial as a prerequisite for extubation to a weaning strategy without a spontaneous breathing trial (direct extubation) in patients with readiness to be weaned criteria and considered at low risk of extubation failure. The main endpoint will be the proportion of patients successfully extubated within the 24 hours after randomization as compared to extubation after a successful spontaneous breathing trial (SBT).

DETAILED DESCRIPTION:
Weaning from mechanical ventilation is a critical step in the course on an ICU stay. Separation from the ventilator should be done at the earliest possible time, but extubation failure is an adverse event that should be avoided. The most common decision-making strategy regarding weaning and extubation is to combine a daily assessment of the patient's "readiness to wean" and a spontaneous breathing trial before to extubate.

The result of the SBT (passed of failed) is often viewed as a "go - no go" indicator of whether or not patients are ready for extubation, but daily practice indicates that the assessment of the SBT is subjective with a frequent natural tendency for clinicians to keep their patients on the 'safe' side, i.e., considering them as not being ready for extubation. However, the results of the SBT should be interpreted based on the pre-test probability. Conducting a SBT in patients while the pre-test probability of success is high will result in false negatives which are likely to delay the decision of extubation. In addition, a pointless SBT may expose patients to anxiety, air hunger and dyspnea which are poorly detected by caregivers. The hypothesis of the present project is that in patients who are at low risk of extubation failure, a SBT is useless and once readiness to wean criteria are met, direct extubation would increase the proportion of patients successfully extubated within the 24 hours after randomization as compared to extubation after a successful SBT.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years and < 65 years old
* Nasal or oral intubation longer than 24 hours and less than 4 days
* Satisfaction to each following weaning readiness criteria:

  1. Respiratory rate < 35 cycles per minute
  2. SpO2 >90% with FiO2<40% and PEEP<8 cmH2O
  3. RASS score between -2 and +2 with low level or no sedatives
  4. No need or low doses of vasopressors
  5. Adequate cough
* Inform consent by patient or legal representative or the close relative or emergency inclusion procedure.

Exclusion Criteria:

* Risk factor for extubation failure as defined by any of the following criteria:

  * Chronic cardiac disease (left ejection fraction below 45%, documented history of cardiogenic pulmonary edema, permanent atrial fibrillation).
  * Chronic respiratory disease (severe COPD, documented restricted lung disease or obesity-hypoventilation syndrome)
  * Body mass index > 30 kg/m2
  * Airway patency problems, including high risk of developing laryngeal edema, inability to deal with respiratory secretions, brain injury, documented swallowing disorders
* Tracheostomy
* Underlying chronic neuromuscular disease
* Do not resuscitate orders
* Pregnant or lacting woman
* Patient under guardianship
* Patient without healthcare insurance
* Refusal to participate and sign the written consent
* Patients with traumatic brain injury
* Post surgery patients
* Patients included in another interventional trial that may have an impact on the evaluation criteria of the present study
* Patient under AME

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-18 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients extubated within the 24 hours after randomization and who will remain free from mechanical ventilation until 72 hours. | From Day 1 to Day 3
  The rate of patients extubated within the 24 hours after randomization and who will remain free from mechanical ventilation until 72 hours.

SECONDARY OUTCOMES:
Occurrence of post extubation acute respiratory failure | Within 28 days after randomization
  Rate of post extubation acute respiratory failure defined by the persistence of more than 30 minutes of at least two predefined criteria
Occurrence of reintubation | Within 28 days after randomization
  Rate of of reintubation with predefined criteria
Unplanned use of non-invasive ventilation or high flow nasal oxygen | Within 28 days after randomization
  Rate of unplanned use of non-invasive ventilation or high flow nasal oxygen
Duration of weaning process from randomization until successful extubation | Within 28 days after randomization
  Number of days from randomization until successful extubation
Total duration of invasive mechanical ventilation from intubation until successful extubation | Within 28 days after randomization
  Total number of days of invasive mechanical ventilation from intubation until successful extubation
Number of Ventilator Free Days between randomization until Day 28 | Within 28 days after randomization
  Number of days without the ventilator and alive from randomization until Day 28
Occurrence of ventilator acquired pneumonia | Within 28 days after randomization
  Ventilator acquired pneumonia will be defined by quantitative distal bronchoalveolar lavage cultures growing ≥104cfu/mL
Length of stay in the ICU and hospital stay | Within 28 days after randomization
  Number of days in the ICU and in the hospital
ICU and hospital mortality | Within 28 days after randomization
  Proportion of patients who died in the ICU and in the hospital
Day 28 mortality | Within 28 days after randomization
  Rate of patients who died at day 28 after randomization
Cumulative incidence of successful extubation over time | Within 28 days after randomization
  Probability of being successfully extubated from randomization until day 28
Duration between randomization and SBT trial | Within 28 days after randomization
  The time between randomization and the onset of the SBT, minutes
Barriers to extubation: logistical, timing, family or patient. | Within 28 days after randomization
  Open
Duration between extubation decision and extubation | Within 28 days after randomization
  Time between extubation decision and extubation, minutes

CONTACTS AND LOCATIONS:
Overall Officials: Martin DRES, Pr, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.